CLINICAL TRIAL: NCT06724731
Title: Role of Combined Ultrasound Elastography in Evaluation the Degree of Liver Fibrosis in Children with Cholesteric Liver Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Mohamed Abdo Hussien, resident doctor at radiology department Faculty of Medicine, Assiut University, Assiut University
Other Study IDs: elastography cholesteric liver
Record Dates: First submitted 2024-11-28; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Liver Diseases
Keywords: liver fibrosis; elastography
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- children patients Cholestatic Liver Disease: evaluate the diagnostic value of the Combi-Elasto technique in assessing liver fibrosis in children with cholestatic liver disease

SUMMARY:
Pediatric CLDs are diverse, encompassing a broad spectrum of conditions, from congenital and metabolic disorders to autoimmune and viral diseases. These chronic liver conditions in children often carry the risk of progressing to fibrosis and cirrhosis. Additionally, certain liver diseases in children exhibit unique characteristics, including varying rates of fibrosis progression. For example, while fibrosis typically takes months to develop in most patients, it progresses much faster in neonates . Approximately 1%-2% of adults, but a significantly higher 17%-30% of children, progress to advanced liver disease and require liver transplantation annually.

the aim of the study to evaluate the diagnostic value of Combi-Elasto technique in detecting degree of liver fibrosis in children with Cholestatic Liver Disease

DETAILED DESCRIPTION:
The prevalence of chronic liver disease (CLD) among children is on the rise globally, driven by various epidemiological shifts, such as the opioid crisis contributing to hepatitis C infections and the obesity epidemic leading to nonalcoholic fatty liver disease (NAFLD) . liver disease affects 1 in every 2,500 infants, and in 2021, children accounted for 13% of all liver transplants in the United States .

Currently, there are no effective pharmacological treatments to prevent or slow the progression of Cholestatic Liver Disease in children. As a result, it is crucial to evaluate the extent of liver fibrosis in children with cholestatic liver disease as early as possible. Early assessment is vital for delaying disease progression, decreasing the need for liver transplantation, and providing essential information for clinical decision-making when transplantation becomes necessary.

Combi-Elasto technique, which integrates elastography with other non-invasive imaging modalities, has emerged as a promising tool for evaluating liver fibrosis. This approach offers several potential benefits, including enhanced diagnostic accuracy, safety, and the ability to assess fibrosis without the need for invasive procedures. Combi-elasto (CE) integrates the benefits of both strain elastography and shear wave elastography. It uses the fibrosis index (FI), activity index (AI), and attenuation coefficient (ATT) to provide precise evaluations of fibrosis levels, inflammation activity, and fatty degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged between 0 and 18 years at the time of enrollment.
* Children must have a confirmed diagnosis of cholestatic liver disease, supported by:

  * Histological confirmation via liver biopsy showing cholestasis.
  * Clinical evidence of cholestasis, such as elevated alkaline phosphatase levels or conjugated hyperbilirubinemia.
* Participants should have a documented history of cholestatic liver disease for at least three months prior to enrollment to ensure that the condition is chronic and allows for adequate assessment of fibrosis progression.

Exclusion Criteria:

* patients without prehepatic ascites
* patients with hepatic space-occupying lesions.
* patients with other serious systemic diseases, such as heart failure, renal failure and mental illness
* patients after liver transplantation.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children patients Cholestatic Liver Disease
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
the accuracy of the Combi-Elasto technique in determining the degree of liver fibrosis in children | baseline
  sensitivity, and specificity of the Combi-Elasto technique in determining the degree of liver fibrosis in children

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhao Y, Wu L, Qin H, Li Q, Shen C, He Y, Yang H. Preoperative combi-elastography for the prediction of early recurrence after curative resection of hepatocellular carcinoma. Clin Imaging. 2021 Nov;79:173-178. doi: 10.1016/j.clinimag.2021.05.020. Epub 2021 May 31. PMID 34087717
- [Background] Lendahl U, Lui VCH, Chung PHY, Tam PKH. Biliary Atresia - emerging diagnostic and therapy opportunities. EBioMedicine. 2021 Dec;74:103689. doi: 10.1016/j.ebiom.2021.103689. Epub 2021 Nov 12. PMID 34781099
- [Background] Zou YG, Wang H, Li WW, Dai DL. Challenges in pediatric inherited/metabolic liver disease: Focus on the disease spectrum, diagnosis and management of relatively common disorders. World J Gastroenterol. 2023 Apr 14;29(14):2114-2126. doi: 10.3748/wjg.v29.i14.2114. PMID 37122598
- [Background] Feldman AG, Sokol RJ. Neonatal cholestasis: emerging molecular diagnostics and potential novel therapeutics. Nat Rev Gastroenterol Hepatol. 2019 Jun;16(6):346-360. doi: 10.1038/s41575-019-0132-z. PMID 30903105